CLINICAL TRIAL: NCT05863936
Title: Clinical Trial of Belimumab Combined With Multi-target Induction Therapy in Adult Patients With Severe Lupus Nephritis
Brief Title: Trial of Belimumab Combined With Multi-target Induction Therapy in Lupus Nephritis
Acronym: BEAM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhi-Hong Liu, MD, Professor in Medicine, Nanjing University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-2023
Record Dates: First submitted 2023-04-19; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Lupus Nephritis; Remission; Safety Issues
Keywords: Lupus nephritis; B cell depletion therapy; Remission
MeSH Terms: conditions — Lupus Nephritis | interventions — belimumab; Immunosuppressive Agents

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Belimumab and multi-target therapy group (Other): Patients with severe lupus nephritis will be enrolled and received pulse methylprednisolone at a dose of 1.5 to 3.0g, followed by intravenous belimumab at a dose of 10mg per kilogram at weeks 2, 4, and 6, and every 4 weeks thereafter. Multitarget therapy will be also administered during the induction phase. Induction therapy will last for 24 weeks.
  Interventions: Drug: Methylprednisolone Injectable Suspension; Drug: Belimumab Injection; Drug: Immunosuppressive Agents

INTERVENTIONS:
Drug: Methylprednisolone Injectable Suspension — Methylprednisolone pulse therapy, total dose from 1500mg to 3000mg.
  Other Names: Methylprednisolone pulse therapy
Drug: Belimumab Injection — Belimumab at a dose of 10mg per kilogram at weeks 2, 4, and 6, and every 4 weeks for 24 weeks.
  Other Names: Beliumab induction therapy
Drug: Immunosuppressive Agents — 1. Mycophenolate Mofetil, oral, 1.0-1.5g per day;
  2. Tacrolimus, oral, 2-4mg per day.
  Other Names: Multi-target immunosuppressive therapy

SUMMARY:
The goal of this single-center, prospective clinical trial is to test the safety and efficacy of belimumab combined with multi-target therapy in the treatment of severe lupus nephritis. The main questions it aims to answer are: lupus nephritis complete remission rate at week 24, and the partial remission rate and safety assessments. Patients with severe lupus nephritis will be enrolled and received pulse methylprednisolone at a dose of 1.5 to 3.0g, followed by intravenous belimumab at a dose of 10mg per kilogram at weeks 2, 4, and 6, and every 4 weeks thereafter. Multitarget therapy will be also administered during the induction phase. Induction therapy will last for 24 weeks. Patients with severe lupus nephritis who only received multi-target therapy during the same period will be enrolled as the control group.

ELIGIBILITY:
Inclusion Criteria:

* Active LN in accordance with the American College of Rheumatology (ACR) diagnostic criteria for SLE (1997), SLE-DAI>10 points (except type Ⅴ LN).
* Patients with active lupus nephritis (type Ⅲ, Ⅳ, Ⅴ, Ⅴ+Ⅲ, Ⅴ+Ⅳ) diagnosed by light microscopy, immunofluorescence microscopy, and electron microscopy according to the ISN/RPS2003 lupus nephritis classification criteria, with pathological chronicity index (CI) less than 3 points and no TMA like changes in interstitial vessels.
* Proteinuria ≥1.5g/24h, with or without active urinary sediment (urinary sediment red blood cell count >100/ul, or white blood cell count >5 /HP, or red blood cell cast, excluding urinary tract infection).
* Serum creatinine <3.0mg/dL or eGFR<30 ml/min/1.73m^2 (CKD-EPI formula).
* Received methylprednisolone pulse therapy within 2 weeks before enrollment, cumulative dose 1.5-3.0g).

Exclusion Criteria:

* Required renal replacement therapy or received renal replacement therapy within 3 months.
* Abnormal liver function with elevated ALT, AST or bilirubin more than 2 times the upper limit of normal.
* Abnormal glucose metabolism, defined as fasting blood glucose concentration ≥7.0mmol/L and/or 2-hour postprandial blood glucose concentration >11.1mmol/L.
* Mycophenolate mofetil, cyclophosphamide, tacrolimus, cyclosporine A, and high-dose intravenous immunoglobulin (IVIG) were used in the past 12 weeks; It did not include oral hormones, azathioprine or tripterygium wilfordii polyglycosides, or intravenous low-dose MP (less than 80mg/ day), or short-term use of cyclosporine A<2 weeks, or leflunomide <4 weeks.
* Known allergy to or contraindication to MMF, tacrolimus, or belimumab; Patients with active infection or intravenous antibiotic use within 1 month before admission.
* Current or past 3 months: active hepatitis B, hepatitis C, tuberculosis, cytomegalovirus pneumonia, active fungal infection, syphilis infection or HIV infection, etc.; Active peptic ulcer; A history of drug use and alcohol abuse; Severe malnutrition (BMI<16 kg/m^2).
* Other active diseases, such as severe life-threatening cardiovascular diseases; Chronic obstructive pulmonary disease, or asthma requiring treatment with oral steroids; Bone marrow suppression caused by SLE activity was excluded: WBC<3000/ul, absolute neutrophil count <1300/ul, and platelet count < 50 000/ul. Patients with active SLE who received double plasma filtration, plasma exchange or high-dose gamma globulin therapy within 4 weeks.
* Patients with malignant hypertension.
* Women who have fertility requirements, refuse contraception or are lactating.
* Other investigators considered that they were not suitable for enrollment and may have rapid disease progression or severe disease complications.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a cumulative complete response at week 24 of treatment. | 24 weeks
  Complete response will be defined as below:
  1. urinary protein less than 0.4g/24h
  2. no active urinary sediment
  3. serum albumin more than 3.5g/dl
  4. and normal SCr.

SECONDARY OUTCOMES:
The proportion of patients with partial response and non-response to treatment. | 24 weeks
  Partial response will be defined as a decrease of more than 50% of the baseline value of urinary protein and less than 3.5g/24h of urinary protein, a decrease of more than 50% of the baseline value of urinary sediment red blood cell count, and a normal or an increase of less than 30% of serum creatinine
Overall response rate at 24 weeks. | 24 weeks
  These will include complete remission and partial remission
Improvement of clinical indicators. | 24 weeks
  Clinical improvement of the disease was assessed using systemic lupus erythematosus disease activity index.
The changes of B cells. | 24 weeks
  The changes of CD20 number in peripheral blood will be observed and investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Hong Liu, MD, Principal Investigator — National Clinical Research Center of Kidney Diseases, Jinling Hospital
Locations (1):
- Jiong Zhang, Nanjing, Jiangsu, China